CLINICAL TRIAL: NCT04169841
Title: Precision Medicine Phase II Study Evaluating the Efficacy of a Double Immunotherapy by Durvalumab and Tremelimumab Combined With Olaparib in Patients With Solid Cancers and Carriers of Homologous Recombination Repair Genes Mutation in Response or Stable After Olaparib Treatment
Brief Title: Study Evaluating the Efficacy of a Double Immunotherapy Combined With Olaparib in Patients With Solid Cancers and Carriers of Homologous Recombination Repair Genes After Olaparib Treatment
Acronym: GUIDE2REPAIR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUIDE2REPAIR
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Immunotherapy
Keywords: immunotherapy; olaparib; durvalumab; tremelimumab; genes mutation
MeSH Terms: interventions — olaparib; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GUIDE2REPAIR patients (Experimental): olaparib + immunotherapy (durvalumab + tremelimumab) during 4 months followed by durvalumab alone as maintenance in patients with solid cancer and in response or stable after prior molecular target therapy by olaparib based on molecular sequencing.
  Interventions: Drug: olaparib, durvalumab, tremelimumab

INTERVENTIONS:
Drug: olaparib, durvalumab, tremelimumab — STEP 1:
  Olaparib 300 mg BID during 8 weeks. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib tablets can be taken with or without food
  STEP 2:
  Olaparib 300 mg during 4 months as per same requirement as below. Durvalumab 1500 mg plus tremelimumab 75 mg via IV infusion Q4W, starting on Week 0, for up to a maximum of 4 doses followed by durvalumab monotherapy 1500 mg via IV infusion Q4W, starting 4 weeks after the last infusion of the combination and in response or stable after prior molecular target therapy by olaparib based on molecular sequencing.

SUMMARY:
The study propose to generate a clinical trial based on precision medicine to evaluate the use of immunotherapy in patients with altered homologous recombination repair genes and without progression after prior targeted therapy.

DETAILED DESCRIPTION:
With the development of cost effective and rapid technology of genome sequencing, precision medicine becomes a new way to think oncology. Current targets involve mainly tyrosine kinase, but DNA repair machinery could also be targetable. Some of DNA repair aberrations have been associated with sensitivity to platinum and poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors like Olaparib, suggesting that treatment with a PARP inhibitor may exploit a synthetic lethal interaction when the presence of alteration of the homologous repair pathway was observed. PARP is involved in multiple aspects of DNA repair, and the PARP inhibitor Olaparib has recently been approved for treating ovarian cancers with BRCA1/2 mutations. In addition, it showed that using a high-throughput, next-generation sequencing assay in prostate cancer, detection of genomic alteration in genes involved in homologous repair pathway BRCA2, ATM, BRCA1, PALB2, CHEK2, FANCA, and HDAC2, is associated with response to olaparib. Thus demonstrating the clinical validation of the usage of precision medicine to position PARP inhibitor like olaparib in different cancer types based on molecular analysis.

Preclinical studies showed DNA damage promotes neoantigen expression. It is possible that increased DNA damage by PARPi would yield greater mutational burden and expand neoantigen expression, leading to greater immune recognition of the tumor. PARPi is also associated with immunomodulation. The PARPi talazoparib increases the number of peritoneal CD8+ T cells and natural killer cells and increases production of interferon (IFN)-γ and tumor necrosis factor-α in a BRCA1-mutated ovarian cancer xenograft model. Hence, addition of PARPi to immune checkpoint blockade could complement the clinical benefit of immune checkpoint inhibition.

Such high level of mutation results in high number of neoantigen and antitumor immune response thus given the rational to use immunotherapy to target such type. A recent paper validate this strategy using the anti PD-1 pembrolizumab Some case reports suggest also that other mutations that induce hypermutated tumor (POLD, POLE, or MYH) could gain benefit from anti PD-1 therapy. Additional DNA repair machinery dysfunction may lead to accumulation of mutations. And such level of mutations could induce better response to immunotherapy. In the lung non-small cell setting high mutation rate were associated with better efficacy of both nivolumab and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria from STEP 1:

1. Capable of giving signed informed consent
2. Exome sequencing of tumor and constitutive DNA should have been already performed
3. Patients must be diagnosed with a solid malignancy with the following cancer histologically confirmed with specified inclusion for each cohort:

   Metastatic breast cancer:

   • In second line

   • third line and after

   Metastatic lung cancer:
   * Non-small cell lung cancer
   * Must have progressed after at least a first line with platinum based therapy

   Metastatic head and Neck cancer

   • Must have progressed after at least a first line with platinum based therapy

   Metastatic endometrial cancer • Progression after 1 prior systemic, platinum-based chemotherapy regimen for EC. Participants may have received up to 1 additional line of platinum-based chemotherapy if given in the neoadjuvant or adjuvant treatment setting. There is no restriction regarding prior hormonal therapy

   Metastatic clear cell renal cancer

   • Must have progressed after at least a line with anti-angiogenic agent. Metastatic pancreatic cancer

   • Must have progressed after at least a line with FOLFIRINOX regimen and/or Gemcitabin based chemotherapy

   Locally advanced or metastatic ovarian cancer

   • Must have received at least one and no more than two lines of prior platinum-containing therapy and progressed after the most recent platinum therapy in a platinum-sensitive timeframe (more than 6 months from the last dose of platinum before randomization)

   Metastatic urothelial cancer • From the second line and regardless previous treatment (except immunotherapy)

   Metastatic prostate cancer
   * Documented evidence of metastatic castration resistant prostate cancer (mCRPC)
   * Ongoing therapy with LHRH analog or bilateral orchiectomy
   * Must have progressed on prior new hormonal agent (enzalutamine or abiraterone) and taxane chemotherapy
4. Presence of mutation in homologous repair gene
5. Age >18 years
6. Performance status ECOG of 0 or 1.
7. Life expectancy ≥ 6 months.
8. At least one lesion measurable as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1)
9. Body weight >30 kg.
10. 10. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential
12. Male patients must use a condom during treatment of STEP1 (olaparib) and STEP2 (durvalumab and tremelimumab) and for 180 days after the last dose when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential
13. Patient is willing and able to comply with the protocol for the duration of the study.
14. For all oral medications patients must be able to comfortably swallow capsules;

Inclusion criteria STEP 2

16. CT Scan evaluation after 6 weeks of olaparib should present response or stable disease as defined by RECIST v1.1 criteria.

Exclusion Criteria:

Exclusion criteria of STEP 1

1. Involvement in the planning and/or conduct of the study
2. Patient with mBRCA1 / 2 that are eligible for current marketing authorization for olaparib (ovarian cancer),and patient eligible for AstraZeneca registration clinical trials, particularly for the prostate cohort
3. Specific exclusion criteria each cohort:

   Metastatic breast cancer:

   • Only for patient second line : patient with mBRCA1 / 2 that are eligible for current marketing authorization for Olaparib (ovarian cancer) and patient eligible for AstraZeneca registration clinical trials).

   Metastatic lung cancer
   * Small cell cancer
   * oncogenic addiction : EGFR mutation or BRAF mutation or ALK rearrangement or ROS1 mutation Locally advanced or metastatic ovarian cancer
   * Patient with mBRCA1 / 2 that are eligible for current marketing authorization for Olaparib (ovarian cancer) and patient eligible for AstraZeneca registration clinical trials.

   Metastatic prostate cancer

   • Untreated or first line patients

   Metastatic head and Neck cancer, Metastatic endometrial cancer, Metastatic clear cell renal cancer, Metastatic pancreatic cancer & Metastatic urothelial cancer:

   • None
4. Participation in another clinical study with an investigational product during within 2 months of first administration of Olaparib.
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
6. Receipt of the last dose of anticancer therapy ≤21 days prior to the first dose of olaparib or 5 times its half-life, whichever is less.
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, ototoxicity, vitiligo, and the laboratory values defined in the inclusion criteria
8. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. Radiotherapy (non-palliative) within 21 days prior the first dose of study drug or within 6 weeks for therapeutic doses of MIBG or craniospinal irradiation. Palliative RT (which would be <30% of the bone marrow) to non-target lesions is allowed.
10. Major surgical procedure within 28 days prior to the first dose of olaparib and patients must have recovered from any effects of any major surgery.
11. Patients unable to swallow orally administered medication and patients with Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs
12. History of allogenic organ, bone marrow or double umbilical cord blood transplantation.
13. Active or prior documented autoimmune or inflammatory disorders
14. Uncontrolled intercurrent illness or patient considered a poor medical risk due to a serious, uncontrolled medical disorder, including but not limited to, ongoing or active infection, symptomatic congestive heart failure
15. Currently taking medications with known risk of prolonging the QT interval or inducing Torsades de Pointes.
16. Concomitant use of known strong or moderate CYP3A inducers.
17. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions or patients with congenital long QT syndrome
18. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
19. History of another primary malignancy
20. History of leptomeningeal carcinomatosis
21. Patient with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of corticosteroids or local CNS-directed therapy to control their CNS disease.
22. History of active primary immunodeficiency
23. Immunocompromised patients
24. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus. Patients with a past or resolved HBV infection are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
25. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab.
26. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
27. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential
28. Prior treatment with any PARP inhibitor including olaparib or immunotherapy.
29. Concomitant use of known strong or moderate cytochrome CYP3A inhibitors and concomitant use of known strong or moderate CYP3A inducers.

    Exclusion criteria of STEP 2

    Patients should not enter the study if any of the exclusion criteria from STEP 1 and the following criteria for STEP 2 are fulfilled:
30. Patient with progression observed on CT scan performed after 6 weeks of olaparib (STEP 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Safety Assessments: progression free survival | 6 months after the initiation of immunotherapy for all cohorts excepted for ovarian cohort where PFS will be evaluated at 12 months.
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: François GHIRINGHELLI, Principal Investigator — Centre Georges Francois Leclerc
Locations (8):
- France (8):
  - CHU Amiens, Amiens
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHU François Mitterrand, Dijon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon

REFERENCES:
- [Derived] Fumet JD, Limagne E, Thibaudin M, Truntzer C, Bertaut A, Rederstorff E, Ghiringhelli F. Precision medicine phase II study evaluating the efficacy of a double immunotherapy by durvalumab and tremelimumab combined with olaparib in patients with solid cancers and carriers of homologous recombination repair genes mutation in response or stable after olaparib treatment. BMC Cancer. 2020 Aug 10;20(1):748. doi: 10.1186/s12885-020-07253-x. PMID 32778095